CLINICAL TRIAL: NCT00157222
Title: Characterizing and Diagnosis's of the Charcot Foot (Charcot Osteoarthropathy) in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: H. Lundbeck A/S (Industry); The Danish Diabetes Association (Other); Clinical and basic research ballerup (Unknown); Steno Diabetes Center Copenhagen (Other)
Other Study IDs: (KF) 01 2587558
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-12-08 (Estimated); Status verified 2005-09

CONDITIONS: Charcot Joint; Diabetic Foot
Keywords: Charcot; Diabetic; osteoporosis
MeSH Terms: conditions — Arthropathy, Neurogenic; Diabetic Foot; Osteoporosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The condition Charcot foot has been known in more than 130 years, and yet there still remains a large effort to find the cause, diagnostic and medical treatment of the condition.

Charcot neuroarthropathy is a progressive disease of bone and joints characterized by often-painless bone and joint destruction in limbs that have lost sensory innervation. The incidence of acute Charcot among diabetic patients is 0,2 % the prevalence is 7,5 %. In the group of patients with neuropathy the prevalence is even higher -29%.

The diagnosis is often made on a clinical basis, particularly in the early stages of the condition. The aim of this study is to find a method that makes the diagnosis primarily on the basis of paraclinical information.

Clinical presentation:

The typical patients have had diabetes in 10 years and have distal symmetrical neuropathy.

The common lesion is unilateral with an acute phase, which may occur either spontaneously or be triggered by a minor trauma. The foot becomes swollen, warm, red and oedematous. Some patients have pain, and the condition could be misdiagnosed as cellulites, acute gout, deep vein thrombosis and osteomyelitis. If the patient has a foot ulcer it is important to rule out osteomyelitis and cellulites.

In the initial phase it is difficult to make the right diagnose because Charcot is a rare condition. This leads to a delay in the treatment of the Charcot foot, which, for the moment, is reduction of weight bearing. The patient is equipped with an air cast, and the non weight-bearing regime is in some cases maintained in 12 months.

The chronic Charcot is characterized by established deformity. The deformity can be in different sites in the foot, the most common is in the mid foot. Because of the deformity there is abnormal weight pressure on the weight bearing sites on the foot. This is associated with callus formation and there is a higher risk for ulceration.

DETAILED DESCRIPTION:
Method:

The investigation is a case control study where the aim is to test a set off clinical tests to see if the diagnose Charcot foot can be made paraclinical. The assumption is, that there are other parameter than the clinical observation that differ between the Charcot patient and a patient with polyneuropathy.

The study will consist of a variety of examinations. All patients will undergo a clinical examination by the same physician, including a neurological status.

The paraclinical examinations consist of blood samples, x-ray of the foot (if normal then MR-scanning of the foot), skeletal Scintigraphy, DEXA scanning, distal blood pressure, beat to beat examination to decide the autonomous neuropathy. If the patient has a positive skeletal scintigraphy and ulceration on the foot, or elevated infection parameter in the blood sample, then a leukocyte scintigraphy will be performed in order to rule out osteomyelitis.

The population that we will include in the study is divided in 5 groups:

1. Patients with diabetes and acute Charcot foot.
2. Patients with diabetes and chronic Charcot foot.
3. Patients with diabetes and amputation of the first toe.
4. Patients with diabetes and polyneuropathy.
5. Patients with diabetes and without polyneuropathy. All patients will undergo the full examination program, with the exception of the cases mentioned above.

Conclusions:

There is need for a better diagnostic of the condition Charcot foot, due to the severe longtime complication in form of disablement. In some cases even amputation of the foot. If the diagnosis is made earlier, obviously one can start the intervention earlier, and this will improve the "survival" of the foot.

Another advantage is that agreed criteria for the diagnosis of Charcot would help in allowing comparison of different treatments.

ELIGIBILITY:
Inclusion Criteria:

* Acute Charcot
* Chronic Charcot
* Polyneuropathy
* Operation of the foot

Exclusion Criteria:

* Pregnancy
* Infection of the foot
* Impert blood flow in the leg.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2005-05; Study Completion 2008-04

CONTACTS AND LOCATIONS:
Overall Officials: Ole L Svendsen, M.D, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark